CLINICAL TRIAL: NCT01439451
Title: Effect of Balance Perturbation to Improve Gait and Balance Control and Prevent Falls in Elderly Persons -A Randomized Control Trial
Brief Title: Effect of Perturbation Training on Balance Control in Elderly Persons
Acronym: BaMPer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Ornit Cohen, IRB Coordinator, Barzilai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BARZI1729
Record Dates: First submitted 2011-09-11; First posted 2011-09-23 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Accidental Falls
Keywords: Balance control; Aging; Balance reactions; Perturbation; above seventy years old

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): perturbation training during walking
  Interventions: Procedure: perturbation training
- controls (Active Comparator): treadmill walking
  Interventions: Procedure: perturbation training

INTERVENTIONS:
Procedure: perturbation training — The experimental and control groups will participate in 3 month training program twice a week 20 minutes each training session
  Other Names: treadmill walking; perturbation training during walking

SUMMARY:
The proposed project is a prospective experimental Randomized Control Trial study design. Independent old adults (age 70 years old and older) who do not suffer from balance problems willing to participate in the study will be tested before and after Peturbation balance training during walking to explore whether there are differences in balance control and balance reactions as a result of training.

DETAILED DESCRIPTION:
A total of 48 old adults will be enrolled, evaluated and trained. They will be randomly assigned to two groups: one exercise group (perturbation training) and one group without perturbation. No gender based differences are expected for the recovery outcome measures so we will be able to pool male and female individuals for this analysis. Each subject of the experimental and of the control groups will be trained on 24 occasions over a period of 10-12 weeks (20-30 minutes, 2-3 times/week). This regimen was based on previous balance training study that demonstrated improvements in balance control with similar training duration and frequency. Gait and balance function and physical activity level will be tested in both groups before, immediately after, 3 and 6 months after completion of the training period to explore the benefit and carryover of training. In addition using monthly phone calls, falls, their severity, functional activity limitations in the home and community setting and health status will be monitored 12 months after the training period.

ELIGIBILITY:
Inclusion Criteria:

* Be 70 years or older, male or female
* Be an independent ambulator (not cane or walker) and provide medical waiver from MD.

Exclusion Criteria:

* Severe focal muscle weakness or paralysis, after Total Hip or knee arthroplasty
* Moderate-severe dementia (Mini-Mental Score < 24).
* Serious visual impairment
* Severe peripheral or compression/entrapment neuropathies.
* Symptomatic orthostatic hypotension, respiratory, cardiovascular, musculoskeletal, or neurological disorders that may interfere with participation in the exercise program.
* Cancer, metastatic or under active treatment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
voluntary and compensatory step execution times in miliseconds | change from baseline to 3 months later
  the time from perturbation to foot contact the floor completing the recovary stepping will be measured in miliseconds

SECONDARY OUTCOMES:
postural sway parameters such as mediolateral sway in milimeters and elliptical area in milimeters squeres | Time 1: pre test' and 3 months later time 2: post testing procedure
  body sway will be measured to evaluate control of posture

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Debi, MD, Study Chair — Barzilai Medical Center
Locations (2):
- Israel (2):
  - Ben-Gurion University of the Negev, Beersheba
  - Beit Yona, Beersheba

REFERENCES:
- [Derived] Batcir S, Shani G, Shapiro A, Alexander N, Melzer I. The kinematics and strategies of recovery steps during lateral losses of balance in standing at different perturbation magnitudes in older adults with varying history of falls. BMC Geriatr. 2020 Jul 20;20(1):249. doi: 10.1186/s12877-020-01650-4. PMID 32689965
- [Derived] Nachmani H, Shani G, Shapiro A, Melzer I. Characteristics of First Recovery Step Response following Unexpected Loss of Balance during Walking: A Dynamic Approach. Gerontology. 2020;66(4):362-370. doi: 10.1159/000505649. Epub 2020 Feb 18. PMID 32069450
- [Derived] Kurz I, Gimmon Y, Shapiro A, Debi R, Snir Y, Melzer I. Unexpected perturbations training improves balance control and voluntary stepping times in older adults - a double blind randomized control trial. BMC Geriatr. 2016 Mar 4;16:58. doi: 10.1186/s12877-016-0223-4. PMID 26944706